CLINICAL TRIAL: NCT06070012
Title: Phase II Open-label, Multi-center Study of Tebentafusp in HLA-A*0201 Positive Previously Untreated Metastatic Uveal Melanoma (mUM) With Integrated Circulating Tumor DNA (ctDNA) Biomarker (TARGET-tebe)
Brief Title: Tebentafusp in HLA-A*0201 Positive Previously Untreated Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Immunocore Ltd (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Associate Professor of Medicine, Hematology/Oncology., University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-165
Record Dates: First submitted 2023-09-20; First posted 2023-10-06 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Uveal Melanoma
Keywords: CD8+ TILs; tumor-associated macrophages (TAMs); PD-L1 (B7- H1); PD-L2 (B7-DC)
MeSH Terms: conditions — Uveal Melanoma | interventions — tebentafusp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tebentafusp (IMCgp100) (Experimental): Dose: 20mcg W1D; 30mcg W2D1; 68mcg W3D1and subsequent doses
  Frequency: Weekly on D1 of 12-week cycles
  Interventions: Drug: Tebentafusp

INTERVENTIONS:
Drug: Tebentafusp — An anti-cancer medication used to treat uveal melanoma. Tebentafusp is a bispecific gp100 peptide-HLA-directed CD3 T cell engager.
  Other Names: Kimmtrak

SUMMARY:
This is a phase II open-label, single-arm, multi-center study of tebentafusp in HLA- A*0201 positive previously untreated (1L) untreated metastatic uveal melanoma (mUM) with an integrated circulating tumor DNA (ctDNA) biomarker.

DETAILED DESCRIPTION:
Uveal Melanoma (UM) is a rare type of melanoma (3.1% of all melanoma incidence, approximately 4000 cases globally per year) with an incidence of 5.3-10.9 cases per million individuals. Despite its rare incidence rate, UM is the most frequent primary intraocular malignancy of the adult eye that affects the vascular layers of the eye (iris, ciliary body, and choroid). UM has a high incidence of metastases, predominantly to the liver, because of the lack of significant lymphatic traffic out of the eye and predominant hematogenous spread.

Tebentafusp has been studied in four clinical studies including IMCgp100-01 (NCT01211262; ≥2L cutaneous and uveal melanoma), IMCgp100-102 (NCT02570308; ≥2L uveal melanoma), IMCgp100-201 (NCT02535078; PD-1 naïve and PD-1 R/R cutaneous melanoma), and IMCgp100-202 (NCT03070392; 1L uveal melanoma vs. physicians' choice chemotherapy). Based on early first-in-human (FIH) studies, tebentafusp 68 mcg was identified as the RP2D; with an intra- patient escalation regimen (20 mcg at C1D1 and 30 mcg at C1D8) and the dose escalated at C1D15. This dose was subsequently evaluated in a recently completed phase -II trial - IMC-p100-202 - that randomized 378 treatment-naïve, HLA-A*0201 positive patients with advanced uveal melanoma on a 2-to-1 ratio to tebentafusp (n = 252) or investigator's choice (IC) of dacarbazine, ipilimumab, or pembrolizumab (n = 126). Based on the data from the IMCgp100-202 study, the current approved dose of tebentafusp is a fixed starting dose of 20mcg (C1D1), followed by 30 mcg (C1D8) and 68mcg at C1D15 and beyond.

ELIGIBILITY:
Inclusion Criteria:

Histologically or cytologically confirmed untreated metastatic uveal melanoma (mUM).

HLA-A*0201 genotype positive as assessed using a CLIA-certified blood typing method and confirmed by central review.

* If HLA-A status is not known, blood for HLA-A testing must be submitted during Screening, and HLA-A*0201 positive status confirmed prior to enrollment using a CLIA- certified blood typing method.
* If the patient is known to be HLA-A*0201 positive, this information must be provided in the Screening packet and centrally reviewed by treating PI and Sponsor-Investigator prior to enrollment.
* The following HLA testing methodologies are suitable to determine HLA-A*0201 positivity:

  * Multiplex real-time PCR based testing performed by entities including but not limited to Labcorp, and American Red Cross.
  * HLA testing as part of peripheral blood molecular profiling technology including but not limited to Caris Life Sciences Molecular Profiling Technology.
* Patients be willing to undergo ctDNA assessment using Signatera assay.
* Have provided newly obtained core biopsy of a tumor lesion not previously irradiated.
* Adequate organ function on screening labs obtained within 4 weeks of Week 1 day 1
* Must meet the following criteria related to prior treatment:

  * No prior systemic therapy in the metastatic or advanced setting including chemotherapy, or targeted therapy.

    * NOTE: Patients must be tebentafusp naïve.
    * NOTE: Patients must not have received prior PD-1, CTLA-4, LAG-3 directed Immune Checkpoint Inhibitor therapy delivered in the adjuvant, and/or neoadjuvant settings unless such therapy was received >6 months prior initial diagnosis of mUM.
  * No prior regional, liver-directed therapy including chemotherapy, radiotherapy, or embolization.
  * Prior surgical resection of oligometastatic disease is allowed.
  * Prior neoadjuvant or adjuvant therapy is allowed provided administered in the curative setting in patients with localized disease.
* Life expectancy of >6 months as estimated by the investigator.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1 at Screening.
* Patients have measurable disease according to RECIST v.1.1.
* All other relevant medical conditions must be well-managed and stable, in the opinion of the investigator, for at least 28 days prior to first administration of study drug.

Exclusion Criteria:

* History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies.
* Clinically significant cardiac disease or impaired cardiac function, including any of the following:

  * Clinically significant and/or uncontrolled heart disease such as congestive heart failure (New York Heart Association grade ≥ 2), uncontrolled hypertension, or clinically significant arrhythmia currently requiring medical treatment.
  * QTcF > 470 msec on screening electrocardiogram (ECG) or congenital long QT syndrome.

    * NOTE: If the initial automated QTcF interval is > 470 msec at screening, for the purpose of determining eligibility, the mean QTcF, based on at least 3 ECGs obtained over a brief time interval (ie, within 30 minutes), should be manually determined by a medically qualified person.
    * NOTE: Acute myocardial infarction or unstable angina pectoris < 6 months prior to Screening.
* Presence of symptomatic or untreated central nervous system (CNS) metastases, or CNS metastases that require doses of corticosteroids within the prior 3 weeks to study Day 1.
* Presence of active brain metastases.

  * NOTE: Patients with brain metastases are eligible if all lesions have been treated surgically and/or radiosurgically and there is no evidence of progression for at least 2 weeks by MRI prior to the first dose of study drug.
  * NOTE: Patients with any evidence of leptomeningeal disease are excluded.
* Active infection requiring systemic antibiotic therapy.

  • NOTE: Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug.
* Known history of uncontrolled active human immunodeficiency virus (HIV), hepatitis B virus (HBV) and/or hepatitis C virus (HCV) infection.

  * NOTE: Testing for HIV, HBV and/or HCV is not necessary unless clinically indicated or the patient has a history of HBV/HCV and/or HIV infection.
  * NOTE: Patients with curatively treated HBV and/or HCV infection may be enrolled. In these instances, HBV (quantitative HBV DNA) and/or HCV (quantitative HCV RNA) resolution must be documented using a quantitative viral load assay.
  * NOTE: Patients with HIV who are stably controlled on highly active antiretroviral therapy (HAART) therapy with a low HIV viral load may be enrolled. In these instances, stable control is defined as HAART compliant with a CD4 count of ≥200 cells/μL, and low viral load is defined as <200 copies/mL on tests done during Screening.
* Malignant disease, other than that being treated in this study. Exceptions to this exclusion include the following:

  * Completely resected carcinoma in situ of any type, resected basal cell and squamous cell carcinomas.
  * Malignancies that were treated curatively and have not recurred within 2 years prior to study treatment;
  * Any malignancy considered to be indolent that has never required therapy Sponsor-Investigator evaluation.
* Any medical condition that would, in the judgment of the Sponsor-Investigator, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results.
* Patients receiving systemic steroid therapy or any other immunosuppressive medication at any dose level, as these may interfere with the mechanism of action of study treatment.

NOTE: Local steroid therapies (eg, otic, ophthalmic, intra-articular or inhaled medications) are acceptable.

* History of symptomatic autoimmune disease including:

  * Interstitial lung disease.
  * Pneumonitis requiring corticosteroid treatment or current pneumonitis.
  * Colitis or inflammatory bowel disease. NOTE: However, patients with a history of autoimmune disease who are currently on physiologic hormone repletion (prednisone or equivalent of 10mg or less) and are otherwise asymptomatic may be enrolled.
* Major surgery within 2 weeks of the first dose of study drug (minimally invasive procedures such as bronchoscopy, tumor biopsy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery and are not exclusionary).
* Radiotherapy within 2 weeks of the first dose of study drug, with the exception of palliative radiotherapy to a limited field, such as for the treatment of bone pain or a focally painful tumor mass.
* Use of hematopoietic colony-stimulating growth factors (eg, G-CSF, GM-CSF, M-CSF) ≤ 2 weeks prior to start of study drug. An erythroid-stimulating agent is allowed as long as it was initiated at least 2 weeks prior to the first dose of study treatment and the patient is not red blood cell transfusion dependent.
* Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation).
* Women of childbearing potential who are sexually active with a non-sterilized male partner, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during study treatment and must agree to continue using such precautions for 6 months after the final dose of investigational product; cessation of birth control after this point should be discussed with a responsible physician.
* Male patients must be surgically sterile or use double barrier contraception methods from enrollment through treatment and for 6 months following administration of the last dose of study drug.
* Receipt of live or attenuated vaccinations 2 weeks prior to starting study therapy. Patients may receive vaccinations on treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA response | At Baseline, at Week 10 of each 12-week cycle, Up to 24 months]
  ctDNA response (defined as ≥0.3 log reduction) in ctDNA-evaluable patients as measured using Signatera assay.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 36 months
  ORR as assessed imRECIST. Percentage of patients with partial response (PR) or complete response (CR) to the treatment. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Overall Survival (OS) | Up to 5 years
  Median length of time from start of treatment that patients remain alive.
1-year Overall Survival (OS) | At one year (post start of treatment)
  The percentage of patients alive at one year after start of treatment.
2-year Overall Survival (OS) | At two years (post start of treatment)
  The percentage of patients alive at two years after start of treatment.
3-year Overall Survival (OS) | At three years (post start of treatment)
  The percentage of patients alive at three years after start of treatment.
Progression-free Survival (PFS) | Up to 5 years
  Median number of months from start of treatment to the date of disease progression or death from any cause. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
6-month Progression-free Survival (PFS) | At 6 months (post start of treatment)
  Percentage of patients without disease progression or death from any cause at six months after start of treatment. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
1-year Progression-free Survival (PFS) | At one year (post start of treatment)
  Percentage of patients without disease progression or death from any cause at one year after start of treatment. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
2-year Progression-free Survival (PFS) | At two years (post start of treatment)
  Percentage of patients without disease progression or death from any cause at two years after start of treatment. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (2):
- United States (2):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No